CLINICAL TRIAL: NCT00881725
Title: A Phase II, Open Label Assessment of Neoadjuvant Intervention With Metformin Against Tumour Expression of Signaling
Brief Title: A Study of Pre-operative Metformin in Prostate Cancer
Acronym: ANIMATE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: University Health Network, Toronto (Other)
Collaborators: Jewish General Hospital (Other)
Responsible Party: Dr. Anthony Joshua, University Health Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMH-ANIMATE-001
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Prostate Cancer
Keywords: Metformin; Prostate Cancer; Radical Prostatectomy; Neoadjuvant Intervention; PTEN/AKT Pathway; Tumour Expression; Ki67 Expression
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): 500mg t.i.d. for 4-12 weeks prior to Radical Prostatectomy
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 500mg tablets t.i.d. for 4-12 weeks prior to Radical Prostatectomy

SUMMARY:
This study will investigate the effect of neoadjuvant metformin therapy in the inhibition of growth and proliferation of prostate cancer cells prior to radical prostatectomy.

DETAILED DESCRIPTION:
Prostate cancer is the most commonly diagnosed malignancy in men in North America, with close to a quarter of a million cases diagnosed in 2007 alone (Joshua et al, 2007). The activation of the PTEN/ AKT pathway is thought to be of importance in prostatic carcinogenesis as it correlates with a poor prognosis (Yoshimoto et al, 2007) (Schmitz et al, 2007). Components of this cellular pathway have pleiotropic targets including the mTOR complex. In model systems, tumours exhibiting activation of PI3K/AKT kinase are sensitive to mTOR inhibitors.

Metformin (1,1-dimethylbiguanide hydrochloride) belongs to the biguanide class of oral hypoglycaemic agents and is a commonly prescribed medication for a number of conditions. It is the first-line drug of choice for the treatment of type 2 diabetes. Its mechanism of action is thought to be the primary inhibition of hepatic glucose output through inhibition of gluconeogenesis. Subsequently, metformin causes a decline in the circulating insulin level (Hundal et al, 2000).

Metformin causes inhibition of the mTOR complex. The mTOR complex is primarily inhibited through activation of AMPK (a component of the PTEN/AKT pathway). Metformin causes reduced hepatic glucose output leading to decreased levels of circulating insulin which causes the secondary inhibition of the mTOR complex. Metformin has also been shown to inhibit cyclin D1 expression and retinoblastoma protein (Rb) phosphorylation. Inhibition of Cyclin D1 and Rb phosphorylation cause inhibition of G1/S phase transition of the cell cycle. This results in the inhibition of cell proliferation (Matsushime et al, 1994).

This study will investigate the effect of neoadjuvant metformin therapy in the inhibition of growth and proliferation of prostate cancer cells prior to radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Patients with histologically confirmed prostate cancer involving at least 20% of at least one unfragmented biopsy core;
2. Over the age of 18 and under the age of 75;
3. Ability to read and understand the consent form, either alone or with the aid of a translator
4. ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%);
5. Patients must have their TRUS biopsy performed at UHN (or at an outside institution if tissue accession can be arranged) in the last 3 months;
6. Patients must have normal organ and marrow function as defined by the following criteria:

   1. Absolute neutrophil count greater than or equal to 1,500/uL
   2. Platelets greater than or equal to 100,000/uL
   3. Total bilirubin less than or equal to 1.5 X institutional ULN
   4. AST(SGOT)/ALT(SGPT) less than or equal to 1.5 X institutional ULN
   5. Creatinine less than or equal to 1.4 X institutional ULN

Exclusion Criteria:

1. Patients who on initial assessment are found to be on treatment with any drug used for the treatment of any form of diabetes, or patients that begin treatment for any form of diabetes during the course of the study;
2. Patients may not be receiving any other investigational, herbal or anticancer agents while on study;
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, congestive heart failure (NYHA Class 3 or greater), cirrhosis with a Child-Pugh level of B or greater or evidence of cardiac dysfunction, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease, clinically significant gastrointestinal conditions (e.g. Crohns disease, ulcerative colitis), COPD or psychiatric illness/social situations that would limit compliance with study requirements;
4. Active malignancy at any other site excluding squamous cell or basal cell carcinomas of the skin
5. Radiotherapy within the past 4 weeks;
6. Patients with a current history of alcohol intake (>2 standard drinks/day) or binge drinking (5 or more drinks (male), or 4 or more drinks (female)) in one session of 1-3 hours;
7. Past history of lactic acidosis or risk factors for lactic acidosis such as congestive heart failure (NYHA Class 3 or greater), hypoxia (resting PO2 < 91%) or renal insufficiency (eGFR < 60 mls/min)
8. Patients taking systemic glucocorticoids or estrogenic compounds.
9. Patients with known hypersensitivity or allergy to metformin or any of its excipients.
10. Patients with a history of impaired liver or kidney function.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Difference in Ki67 staining | Pre-Surgery

SECONDARY OUTCOMES:
Other immunohistochemical assays: IR, IGF-1R, p70S6K, AMPK, MVD, Cleaved caspase 3, PTEN, c-Myc | Pre-Surgery
Differences in measures of insulin resistance: waist/hip ratio, fasting blood glucose, post-prandial blood glucose, weight | Pre-Surgery, Post-Surgery
Differences in PSA levels | Pre-Surgery, Post-Surgery
Incidence of adverse events, serious adverse events, and grade 3-4 toxicities | Pre-Surgery, Post-Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, M.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Joshua AM, Evans A, Van der Kwast T, Zielenska M, Meeker AK, Chinnaiyan A, Squire JA. Prostatic preneoplasia and beyond. Biochim Biophys Acta. 2008 Apr;1785(2):156-81. doi: 10.1016/j.bbcan.2007.12.001. Epub 2007 Dec 8. PMID 18166163
- [Background] Yoshimoto M, Cunha IW, Coudry RA, Fonseca FP, Torres CH, Soares FA, Squire JA. FISH analysis of 107 prostate cancers shows that PTEN genomic deletion is associated with poor clinical outcome. Br J Cancer. 2007 Sep 3;97(5):678-85. doi: 10.1038/sj.bjc.6603924. Epub 2007 Aug 14. PMID 17700571
- [Background] Schmitz M, Grignard G, Margue C, Dippel W, Capesius C, Mossong J, Nathan M, Giacchi S, Scheiden R, Kieffer N. Complete loss of PTEN expression as a possible early prognostic marker for prostate cancer metastasis. Int J Cancer. 2007 Mar 15;120(6):1284-92. doi: 10.1002/ijc.22359. PMID 17163422
- [Background] Hundal RS, Krssak M, Dufour S, Laurent D, Lebon V, Chandramouli V, Inzucchi SE, Schumann WC, Petersen KF, Landau BR, Shulman GI. Mechanism by which metformin reduces glucose production in type 2 diabetes. Diabetes. 2000 Dec;49(12):2063-9. doi: 10.2337/diabetes.49.12.2063. PMID 11118008
- [Background] Matsushime H, Quelle DE, Shurtleff SA, Shibuya M, Sherr CJ, Kato JY. D-type cyclin-dependent kinase activity in mammalian cells. Mol Cell Biol. 1994 Mar;14(3):2066-76. doi: 10.1128/mcb.14.3.2066-2076.1994. PMID 8114738